CLINICAL TRIAL: NCT05736289
Title: Evaluation of Mitral Valve Insufficiency Under General Anesthesia
Acronym: MITIGATE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Denise P. Veelo, Principal Investigator, Associate Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W22_423
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Mitral Regurgitation; Mitral Valve Disease; Mitral Valve Insufficiency
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Percutaneous mitral valve repair: Patients undergoing percutaneous mitral valve repair under general anesthesia for mitral valve regurgitation.
- Surgical mitral valve repair or replacement: Patients undergoing surgical mitral valve repair or replacement for mitral valve regurgitation.

SUMMARY:
Observational study in adult humans undergoing surgical or cardiological intervention for mitral valve insufficiency. Investigators aim to evaluate hemodynamic changes on an arterial pressure waveform level in patients before and after mitral valve intervention using Nexfin (BMEYE, Amsterdam, the Netherlands) continuous non-invasive hemodynamic monitoring, using finger cuff based technology to register beat-to-beat data

ELIGIBILITY:
Inclusion Criteria:

* All patients with moderate or severe mitral valve insufficiency undergoing cardiothoracic surgery or percutaneous treatment for this condition
* Adult patients (>18 years)

Exclusion Criteria:

* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate or severe mitral valve insufficiency undergoing cardiothoracic surgery or percutaneous treatment for their mitral valve condition.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Arterial pressure waveform changes | Before and during general anesthesia for mitral valve repair or replacement, ranging from 1 to 5 hours.
  Arterial pressure waveform as recorded by a continuous non invasive hemodynamic monitoring system.

CONTACTS AND LOCATIONS:
Overall Officials: Denise P Veelo, MD PhD, Principal Investigator — Amsterdam University Medical Center - University of Amsterdam
Locations (1):
- Amsterdam University Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
none as of writing